CLINICAL TRIAL: NCT06602960
Title: Nextsense Brain-sensing Buds Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped due to technical difficulties in verifying participants' receipt of the intervention-specifically, whether they opened the intervention message.We completed a preliminary analysis of data from 40 participants.
Sponsor: NextSense, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Sterling IRB #12205
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Sleep; Sleep Quality; Sleepiness, Daytime; Technology
Keywords: sleep; mindset about sleep; brain-sensing buds
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (Active Comparator): All arms receive identical instructions during the onboarding session, which includes information about the study's purpose and the use of Fitbit and NextSense brain-sensing earbuds. Participants are provided with a Fitbit and NextSense brain-sensing earbuds upon enrollment in the study and are instructed to wear them during weeks 3-4. Throughout the 4 weeks, participants complete short daily surveys and longer weekly surveys. At the end of the study, participants complete an "offboarding" survey.
  In this arm, participants will receive accurate feedback about their sleep data.
  Interventions: Behavioral: Accurate Sleep Data Feedback
- Intervention Group 1 (Experimental): All arms receive identical instructions during the onboarding session, which includes information about the study's purpose and the use of Fitbit and NextSense brain-sensing earbuds. Participants are provided with a Fitbit and NextSense brain-sensing earbuds upon enrollment in the study and are instructed to wear them during weeks 3-4. Throughout the 4 weeks, participants complete short daily surveys and longer weekly surveys. At the end of the study, participants complete an "offboarding" survey.
  In this arm, participants will receive inflated feedback about their sleep data, suggesting better sleep quality than detected by Fitbit (actual sleep hours +10%).
  Interventions: Behavioral: Inflated Sleep Data Feedback
- Intervention Group 2 (Experimental): All arms receive identical instructions during the onboarding session, which includes information about the study's purpose and the use of Fitbit and NextSense brain-sensing earbuds. Participants are provided with a Fitbit and NextSense brain-sensing earbuds upon enrollment in the study and are instructed to wear them during weeks 3-4. Throughout the 4 weeks, participants complete short daily surveys and longer weekly surveys. At the end of the study, participants complete an "offboarding" survey.
  In this arm, participants will receive deflated feedback about their sleep data, suggesting poorer sleep quality than detected by Fitbit (actual sleep hours -10%).
  Interventions: Behavioral: Deflated Sleep Data Feedback
- Intervention Group 3 (Experimental): All arms receive identical instructions during the onboarding session, which includes information about the study's purpose and the use of Fitbit and NextSense brain-sensing earbuds. Participants are provided with a Fitbit and NextSense brain-sensing earbuds upon enrollment in the study and are instructed to wear them during weeks 3-4. Throughout the 4 weeks, participants complete short daily surveys and longer weekly surveys. At the end of the study, participants complete an "offboarding" survey.
  In this arm, participants will receive accurate feedback about their sleep data along with sleep-related educational information.
  Interventions: Behavioral: Accurate Sleep Data Feedback + Sleep-related Educational Information

INTERVENTIONS:
Behavioral: Accurate Sleep Data Feedback — Participants will receive accurate feedback about their sleep data.
  Arms: Control Group
Behavioral: Inflated Sleep Data Feedback — Participants will receive inflated feedback about their sleep data, suggesting better sleep quality than detected by Fitbit (actual sleep hours +10%).
  Arms: Intervention Group 1
Behavioral: Deflated Sleep Data Feedback — Participants will receive deflated feedback about their sleep data, suggesting poorer sleep quality than detected by Fitbit (actual sleep hours -10%).
  Arms: Intervention Group 2
Behavioral: Accurate Sleep Data Feedback + Sleep-related Educational Information — Participants will receive accurate feedback about their sleep data along with sleep-related educational information.
  Arms: Intervention Group 3

SUMMARY:
The purpose of this clinical trial is to explore how the presentation of sleep data impacts sleep quality, sleep-related behaviors (such as sleepiness), and sleep-related anxiety and stress. The study aims to answer the following key questions:

1. Does receiving sleep-related feedback from a wearable sleep tracker affect an individual's mindset about sleep?
2. How does the mindset about sleep influence sleep quality, sleepiness, and stress/anxiety levels related to sleep?
3. Does the feedback on sleep data moderate the relationship between one's mindset about sleep and their sleep quality?

Participants will:

1. Be randomly assigned to receive different types of feedback about their sleep data to determine if the way sleep data is presented influences self-reported sleep quality, sleepiness, and sleep-related stress.
2. During the baseline period (Weeks 1-2), complete daily and weekly surveys assessing their sleep habits, beliefs about sleep, anxiety, stress, and mindset regarding sleep.
3. For Weeks 3-4, wear a Fitbit and Brain-Sensing earbuds, receiving daily feedback on their sleep.
4. At the end of the study, provide feedback on their experience using the devices. Participants may choose to return the devices or keep them after the study concludes.

DETAILED DESCRIPTION:
With the growing prevalence of sleep-tracking wearables available to consumers, understanding the psychological and behavioral impacts they have on users is important. Recent advancements in wearable technology allow for monitoring various sleep parameters, providing users with extensive data on their sleep patterns. The study aims to examine how the presentation of sleep data influences user sleep quality, sleep-related behaviors, including sleepiness, and sleep-related anxiety and stress. It will evaluate how the presentation of sleep data affects individuals' perceptions of sleep and related health issues, including daytime sleepiness and perceived sleep quality. Participants will receive sleep data feedback based on new methods assessed using Fitbit, brain-sensing earbuds, and other factors that might impact sleep. Additionally, the study seeks to offer valuable insights into sleep research, behavioral psychology, and wearable technology.

ELIGIBILITY:
Inclusion Criteria:

* All participants have the capacity to understand the informed consent for study participation and ability for subject to comply with the requirements of the study
* Experiencing mild to moderate sleep disturbances, but without sleep disorder diagnosis
* Naïve to sleep tracker use
* Age 25-65

Exclusion Criteria:

* Participants who have used any type of sleep tracker, such as Oura, Fitbit, Google Fit, Garmin Connect, or Apple Watch Sleep
* Health conditions (i.e., cancer, cognitive impairment, panic disorder, post-traumatic stress disorder, sleep apnea, insomnia, restless leg syndrome, Parkinson's disease)
* Use of Modafinil (Provigil), Methylphenidate (Ritalin), Sodium oxybate (Xyrem), Melatonin, Benadryl, Wakix, Sunosi or prescription medications for ADHD Enrollment in other sleep studies
* Women who are pregnant or who are currently nursing/breastfeeding will be excluded from this study.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Participant-reported Sleep Quality | 4 weeks (Week 1 - Week 4): measured at baseline, in daily surveys.
  Measured via self-report using the 15-item Groningen Sleep Quality Scale, with scores ranging from 1 to 14. A score of 14 indicates poor sleep quality the previous night.
Sleep data - Total hours of sleep | 2 weeks (Week 3 - Week 4): measured daily, sleep data tracked by Fitbit will be transmitted to the Alethios platform automatically once a day.
  Total hours of sleep data tracked by Fitbit
Modified Karolinska Sleepiness Scale | 4 weeks (Week 1 - Week 4): measured at baseline, in daily surveys.
  Sleepiness, measured via self-report using the 1-item modified Karolinska Sleepiness Scale, ranges from 1 to 10, with 1 indicating extreme alertness, 3 alert, 5 neither alert nor sleepy, 7 sleepy but no difficulty remaining awake, 9 extremely sleepy, fighting sleep, and 10 extremely sleepy, falling asleep all the time.
Fitbit tracked Sleep Quality | 2 weeks (Week 3 - Week 4): measured daily, sleep data tracked by Fitbit will be transmitted to the Alethios platform automatically once a day.
  Fitbit sleep score, ranging from 0 to 100, indicates sleep quality: 90-100 is excellent, 80-89 good, 60-79 fair, and 0-59 poor, based on duration, disturbances, and restorative sleep.

SECONDARY OUTCOMES:
Anxiety, Stress, and Mindset related to Sleep | 4 weeks (Week 1 - Week 4): measured at baseline, in weekly surveys.
  Measured via self-report using the 7-item survey.
Dysfunctional Beliefs and Attitudes about Sleep 16-item | 4 weeks (Week 1 - Week 4): measured at baseline, in weekly surveys.
  Sleep-related mindset, measured via self-report using the 16-item Dysfunctional Beliefs and Attitudes about Sleep, involves calculating the average of the scores from all 16 items. Higher average scores indicate a stronger endorsement of sleep-disruptive beliefs, which are considered maladaptive.
Modified Insomnia Severity Index | Week 2 and Week 4: measured twice.
  Severity of Sleep Problems, measured via self-report using the 5-item Insomnia Severity Index, modified to replace Insomnia with Sleep.
Satisfaction with sleep | Week 2 and Week 4: measured twice.
  Measured via self-report using a single item, with scores ranging from 1 to 5, where 1 indicates very satisfied and 5 indicates very dissatisfied.
Sleep Problems Interference with Daily Functioning | Week 2 and Week 4: measured twice.
  Measured via self-report using a single item, with scores ranging from 1 to 5, where 1 indicates not at all interfering and 5 indicates very much interfering.
Pre-Sleep Arousal Scale | 4 weeks (Week 1 - Week 4): measured at baseline, in weekly surveys.
  Pre-sleep arousal, measured via self-report using the 16-item Pre-Sleep Arousal Scale, with items rated on a 5-point Likert scale from 1 (not at all) to 5 (extremely). The sum of scores from the first 8 items reflects somatic pre-sleep arousal, and the sum of scores from the last 8 items reflects cognitive pre-sleep arousal. Clinically relevant cut-off scores will be used: ≥14 for somatic pre-sleep arousal and ≥20 for cognitive pre-sleep arousal.

OTHER OUTCOMES:
Virtual Research Participation | Once at the end of the study, through study completion, which averages approximately 1 year.
  Measured via self-report using the 10-item questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Mi Kim, PhD, Principal Investigator — MandK Consulting Partners; Michele D Nelson, PhD, Principal Investigator — MandK Consulting Partners
Locations (1):
- Alethios (Virtual Study Platform), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No